CLINICAL TRIAL: NCT04521985
Title: The Effectiveness of Gastroesophageal Reflux Improvement in Different Treatments in Thoracolumbar Kyphotic Patients Who Fulfill the Surgical Indications
Brief Title: Thorcolumbar Kyphosis Patients With GERD
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006117RINB
Record Dates: First submitted 2020-08-16; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: the GERD Occurence
Keywords: thoracolumbar kyphosis; esophageal motility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thoracolumbar kyphosis: patients undergoing thoracolumbar kyphosis surgery
  Interventions: Procedure: thoracolumbar kyphosis surgery

INTERVENTIONS:
Procedure: thoracolumbar kyphosis surgery — patients receiving surgery or not

SUMMARY:
The investigator aimed to investigate the gastroesophageal reflux disease (GERD) along with esophageal motility in thoracolumbar kyphotic patients who meet surgical spinal correction criteria. Because some patients refused to receive spinal correction surgery, our patients divided into surgical and non-surgical treatment (for example: brace) groups. The investigator intended to use (1) multichannel intraluminal impedance-pH (MII-pH) monitoring to assess the height, non-acidic and acidic regurgitation of gastroesophageal reflux disease (GERD) (2) high resolution impedance manometry (HRIM) to esophageal motility between pretreatment and posttreatment period. (3) the questionnaire to evaluate the reflux-related symptoms: the frequency scale for the symptoms of GERD (FSSG), gastrointestinal symptom rating scale (GSRS) and Carlsson-Dent self-administered questionnaire (QUEST)

DETAILED DESCRIPTION:
Background: the investigator aimed to investigate the gastroesophageal reflux disease (GERD) along with esophageal motility in thoracolumbar kyphotic patients who meet surgical spinal correction criteria. Because some patients refused to receive spinal correction surgery, our patients divided into surgical and non-surgical treatment (for example: brace) groups. The investigator intended to use (1) multichannel intraluminal impedance-pH (MII-pH) monitoring to assess the height, non-acidic and acidic regurgitation of gastroesophageal reflux disease (GERD) (2) high resolution impedance manometry (HRIM) to esophageal motility between pretreatment and posttreatment period. (3) the questionnaire to evaluate the reflux-related symptoms: the frequency scale for the symptoms of GERD (FSSG), gastrointestinal symptom rating scale (GSRS) and Carlsson-Dent self-administered questionnaire (QUEST)

Objectives:

1. To determine whether acid or weakly acidic reflux in to the esophagus decreases after patients receiving treatment.
2. To investigate the change of esophageal motility after patients receiving treatment.
3. To determine whether the GERD symptoms would get improved after surgical or nonsurgical treatment.

Patients and methods: After the surgeon explained the spinal correction surgery, patients decided to recieve the correction surgery or wear brace treatment. Three types of evaluation were conducted in (1) patients receiving surgical correction [preoeprative and postoeprative surgical spinal correction (within 6 months)] (2) patients receiving brace treatment for 3 month [pretreament and wearing brace after 3 month within 6 months]; namely, HRIM, 24h MII-pH monitoring and three different questionniare surveys: the freqeuncy scale for the symptoms of GERD (FSSG), gastrointestinal symptom rating scale (GSRS) and Carlsson-Dent self administered questionniare (QUEST).The primary outcome was to evaluate the efficacy of surgical spinal correction for GERD by questionniare in patients with severe kyphotic deformity.

Expected result: 1.To precisely estimate efficacy of kyphosis surgical correction and brace treatment 2. To determine whether spinal correction for kyphosis patients with GERD is a surgical indication for the treatment of GERD along with for the treatment of kyphotic deformity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with thoracolumbar kyphotic deformity meet the surgical correction indication. These thoracolumbar kyphotic deformity caused by osteoporossis, multiple vertebral fractures, adult idiopathic scoliosis, camptocormia as a result of Parkinson's disease, degenrative de novo kyphoscoliosis or

Exclusion Criteria:

* Age less than 20 year old
* Previous history of abdominal operation, including the esophagus and stomach.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will fulfill the surgical criteria of thoracolumbar correction surgery.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
GERD occurrence | GERD occurence change from pre-treatment and after receiving treatent within 6 months
  patients wiht GERD symptoms

IPD SHARING:
Plan to Share IPD: No
due to ethical problem